CLINICAL TRIAL: NCT06570499
Title: Precision, Patient Satisfaction and Timing of Complete-arch Digital Implant Impression With a Conventional Impression, an Intraoral Scanner and a Photogrammetry Technique: A Prospective Clinical Comparative Study
Brief Title: Comparison of Conventional Impressions, Intraoral Scanners and Digital Photogrammetry for Full-arch Implant Prosthesis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Nathalie Robert, Phd student, Centre Hospitalier Universitaire de Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: B7072024000032
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Dental Implant Failed
Keywords: accuracy, photogrammetry, dental implant

STUDY DESIGN:
Intervention Model Description: a group of patients: 6 different impressions taken from the same patient. Analysis of the impressions in a second step
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with 4-8 osseointegrated implants (Other): On the patient, we will successively take 6 impressions (2 conventional, 2 intraoral scanner, 2 photogrammetry) and then analyze these impressions to measure the repeatability of a technique. After each type of impression, a satisfaction questionnaire in VAS format will be given to the patient.
  Interventions: Other: Implant impression

INTERVENTIONS:
Other: Implant impression — definitive impressions on implants

SUMMARY:
The aim of this clinical trial is to compare implant-supported definitive impressions in edentulous patients (mandible or maxilla) with 4 to 8 osseointegrated implants. The main questions it aims to answer are :

The primary outcome of this prospective clinical comparative study is to analyse the precision of a complete-arch impression.

The secondary aim is to obtain patient satisfaction with these new types of impression.

The different impressions (conventional, intraoral scanner and photogrammetry) will be taken twice on the same patient.

DETAILED DESCRIPTION:
For each patient, 6 impressions were taken in the same order: 2 IOS, 2 photogrammetry, 2 conventional impressions. A satisfaction questionnaire in the form of a Visual Analogue Scale (VAS) was given after each group of impressions. The time required for each impression was also measured

Clinical and laboratory Protocol The conventional impression will taken in plaster using an open tray technique (Dr. Balzer® Special plaster, Siladent). The impression copings (Impression Coping Open Tray Multi-unit, NobelBiocare) will be screwed onto the transgingival abutments. The plaster wil then prepared with the 50:100 water/powder ratio recommended by the manufacturer. The resulting impression will then cast with low-extension plaster and digitized using a high-precision laboratory scanner. The entire procedure wil be conducted twice.

The IOS impression will obtained using an intraoral scanner (TRIOS4; 3Shape A/S) with implant scan bodies screwed at the multiunit abutment level (Elos Accurate Multi-Unit; Elos Medtech). The IOS device will be a wireless, powder-free scanner with a pen grip, based on confocal microscopy laser technology, and operated with software version 1.4.7.5, calibrated immediately before the impression. The scanning strategy will be consistent for all procedures, consisting of a first scan of the gingiva and implants, in accordance with the manufacturer's recommendations. The scanbodies will be then hand screwed and a second scan will be performed using the following scan path: from the last distal implant in a zigzag pattern[26]. The entire procedure will be conducted twice.

Photogrammetry will be carried out using an Imetric camera (ICam4D; Imetric4D Imaging Sàrl). The first step will be to use an intraoral scanner to scan the gingiva and optical markers screwed onto the transgingival abutments. In a second step, the scan bodies with superﬁcial target points and titanium interfaces (ICamBody; Imetric4D Imaging Sàrl) will be hand screwed to the transgingival components. The ICamBodies will be placed with a visible edge in accordance with the manufacturer's recommendations. The operator will set up the photogrammetric camera (ICam4D; Imetric4D Imaging Sàrl) and directly capture the scan bodies from right to left at 10 cm to 15 cm from the lips. At least 2 sides of the scan body, with 3 target points on each side, will be captured according to the manufacturer's instructions. The scanbodies will be unscrewed and screwed back in random order and a second recording will be made after recalibrating the photogrammetry. The coordinates from the photogrammetry will be exported the to dedicated software to be merged with the STL file form the intraoral scanner. The entire procedure will be conducted twice.

Patient-reported outcome measures (PROMs) PROMs will be obtained using a Visual Analog Scale (VAS, [27]) immediately after the impression. For each impression technique, six domains will be used to evaluate which of the two was less unpleasant: (a) opinion on treatment length (1 = unsatisfactory to 10 = excellent), (b) comfort level during impression procedures (1 = unsatisfactory to 10 = excellent), (c) anxiety level before impression procedures (1 = high to 10 = low), (d) unpleasant taste during/after impression procedures (1 = bad taste to 10 = none), (e) nausea during the impression procedure (1 = severe to 10 = none), and (f) pain during impression procedures (1 = painful to 10 = none). For all Visual Analog Scales (VAS), higher scores indicated greater satisfaction with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* edentulous maxilla or mandible with 4 to 8 osseointegrated implants (NobelBiocare®) and transgingival abutments tightened to 35N/cm (Multi-unit, NobelBiocare®).

Exclusion Criteria:

* Patients with non-osseointegrated implants
* Patients with different implant systems
* Patients with incomplete edentulism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Compare the precision of a complete-arch impression | The impressions will be taken on the same day, the appointment lasts one hour.
  6 impressions are taken on one patient

SECONDARY OUTCOMES:
Obtain patient satisfaction with these new types of impression. | The questionnaire is handed out after the impressions, during the only appointment of this study (one hour).
  Patients complete a satisfaction questionnaire in VAS format

CONTACTS AND LOCATIONS:
Overall Officials: Marc Pr Lamy, Phd, Study Director — Centre Hospitalier Universitaire de Liege
Locations (1):
- Institut de Dentisterie, Liège, Liege, Belgium

IPD SHARING:
Plan to Share IPD: No